CLINICAL TRIAL: NCT02228421
Title: A Phase IV Multicenter Trial to Evaluate Real-world Pharmacoeconomics of Crizotinib and Its Companion Diagnostic Test in Advanced ALK-positive Non-small Cell Lung Cancer (NSCLC) Patients
Brief Title: Study to Evaluate Real-world Pharmacoeconomics of Crizotinib in NSCLC Patients
Status: Terminated | Type: Observational
Sponsor: PeriPharm (Other)
Collaborators: Personalized Medicine Partnership for Cancer (Other); Jewish General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PMPC-03
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2016-10

CONDITIONS: Non-small Cell Lung Cancer Metastatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a phase IV multicenter trial to evaluate the pharmacoeconomic (PE) impact of crizotinib and its companion diagnostic test used in a real-life setting in advanced ALK-positive non-small cell lung cancer (NSCLC) patients.

NSCLC represent 80% of all new cases of lung cancer. One molecular subtype of NSCLC is the ALK-positive subtype. The anaplastic lymphoma kinase (ALK) is a transmembrane receptor tyrosine kinase. Activation of ALK occurs through the formation of gene fusions and in NSCLC, the gene fusion partner for ALK is primarily EML4. The resulting fusion protein is capable of activating the ALK kinase domain, leading to cell growth. The estimated prevalence for ALK rearrangements in NSCLC is 3-5%, and is more commonly found amongst patients with adenocarcinoma histology, in never smokers and in those who are known to be wild type for EGFR and KRAS.

Crizotinib is a potent inhibitor of ALK and is approved for the treatment of advanced ALK+ NSCLC patients. This is an example of personalized medicine, where patients are selected for treatment based upon a molecular assay, and are provided a specific therapy (crizotinib) for their disease. The pharmacoeconomic impact of using genetic information in early treatment decisions in NSCLC has not been determined.

The study will enable real-life Heath Economics and Outcome Research (HEOR).

Approximately 90 patients will be recruited. Patients will be asked to complete quality-of-life questionnaires at regular intervals in a real-life setting of treatment with crizotinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed locally advanced or metastatic NSCLC
* Presence of the ALK-fusion oncogene (ALK+) as determined using a validated testing platform
* Planned first or second-line treatment with crizotinib
* Signed and dated IRB-approved informed consent document
* Ability to read and understand English or French
* 18 years of age or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) found positive for ALK mutation.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2015-02; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
The pharmacoeconomic impact of using personalized medicine for the treatment of ALK+ lung cancer. | From the date of registration until date of death from any cause, assessed up to 60 months.
  Pharmacoeconomic impact (cost-effectiveness and cost utility) will be evaluated by questionnaires completed by the patient and caregiver. These include quality of life, health resource utilization, work productivity and activity impairment, and health questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Agulnik, MD, Principal Investigator — Jewish General Hospital; Victor Cohen, MD, Principal Investigator — Jewish General Hospital
Locations (3):
- Canada (3):
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CSSS de Rimouski-Neigette, Rimouski, Quebec